Throwers Ten Exercises On Upper Extremity Function and Explosive Power in Wheelchair Basketball and Basketball Players

NCT Number: 04019990

Date of the document: 20.11.2019

**Objective:** The purpose of this study was to investigate the effect of Thrower's Ten Exercise program which has impressive results in upper extremity sports in wheelchair basketball and basketball players. Twelve male wheelchair basketball players with average of  $35,6\pm10,9$  years and twelve male basketball players with average of  $28,9\pm7,2$  years were included in the study.

**Design:** Cross-sectional study.

**Method:** J-Tech medical tracker freedom was used for measuring upper extremity muscle power and range of motion. Medicine ball throw test was used for plyometric power. Athletes were involved in 8 weeks Thrower's Ten exercise program. After 8. Weeks and 12. Weeks assessments were repeated.

**Statistical Analysis Plan:** The data was analyzed using SPSS software version SPSS 21 (IBM Inc., Armonk, NY, USA). Type 1 error was set 5% and 95% confidence interval was used for all analysis. Numerical data was shown with mean and standard deviation. To determine between group differences in independent groups Mann-Whitney-U test was used. Benferroni correction was used for non-parametric post-hoc analysis. In order to analyze within group changes Friedman non parametric analysis of variance was used. To determine the statistically significant differences occurred between two dependent groups Wilcoxon test was used for post-hoc analysis.